CLINICAL TRIAL: NCT00304148
Title: Prospective Cohort Study of Chronic Renal Insufficiency
Brief Title: SDCC - Prospective Cohort Study of Chronic Renal Insufficiency
Acronym: CRIC
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Johns Hopkins University (Other); Case Western Reserve University (Other); University of Michigan (Other); University of Illinois at Chicago (Other); Tulane University (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: DK60990; U01DK060990 (NIH)
Record Dates: First submitted 2006-03-14; First posted 2006-03-17 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Renal Insufficiency Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, urine, serum, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CRIC Cohort
- CRIC Subcohort

SUMMARY:
Chronic kidney disease (CKD) is a silent epidemic affecting more than 37 million Americans. The burden of morbidity and mortality associated with CKD derives from its frequent progression to end-stage kidney disease (ESKD) and the disproportionate risk of cardiovascular disease (CVD) and associated complications. CKD is strongly and independently associated with CVD, even after adjustment for traditional CVD risk factors. This led to the hypothesis that other risk factors augment the rate of CVD in the setting of CKD. Hence, many patients with progressive renal disease succumb to fatal CVD events before they need renal replacement therapy.

The National Institute of Diabetes, Digestive, and Kidney Diseases (NIDDK) established the Chronic Renal Insufficiency Cohort (CRIC) Study in 2001 with the initial goal of elucidating the relationship between CKD and CVD. Since its inception, the CRIC Study has recruited and followed a racially and ethnically diverse cohort of over 5,000 participants with reduced kidney function from 13 clinical recruitment sites across the US. The original aim of CRIC was to establish a clinical research laboratory designed to (a) identify novel predictors of CKD progression, and (b) characterize the manifestations of CVD and identify its risk factors among individuals with CKD. The CRIC Study has examined a broad set of etiological factors (clinical, behavioral, and biomarker-associated) potentially responsible for both progressive CKD and CKD-related morbidities, especially those early in the course of CKD. Characterizing relationships between these risk factors and outcomes should facilitate identification of high-risk subgroups with CKD and guide enrollment into preventive treatment trials and application of preventive therapies. Over time, the scientific focus and the CRIC investigator network have broadened extensively through a highly successful ancillary studies program that has included more than 100 projects, most of which have been funded through federal grants. To date, the CRIC Study's investigative activities have resulted in over 300 published scientific papers with many additional manuscripts in development.

DETAILED DESCRIPTION:
Study Visits and Participant Contact

During its 5th and final phase, the 7 Clinical Centers comprised of 12 sites will extend participant follow-up for participants who have not reached ESKD before the inception of Phase 5 by conducting 2 study visits. For all participants, Visit 1 is conducted in person at the study site. Visit 2 can be conducted in person or by telephone. For participants who enrolled in one or more Phase 4 subprotocols, Visit 2 requires a blood draw for a creatinine measurement. The blood draw can be performed at the study site, at a commercial laboratory, or at the participant's home. The principal focus for these study visits is to ascertain kidney and clinical CVD outcomes, both of which are of particular importance for the participants who enrolled in the three Phase 4 subprotocols. Participants may be contacted at other times during the year to answer additional questions or to join ancillary studies. Participants who are known by the study team to have ESKD will not have any in-person visits or scheduled telephone calls.

Phase 5 Visit 1

Participants without ESKD will complete one initial visit through the end of 2024 (Visit 1) and one follow up visit during the following year (Visit 2). Data collection has been streamlined in accordance with the Phase 5 objectives . At the in-person visit, informed consent will be obtained for continued participation in the CRIC Study. Blood pressure, weight, and medical history data will be obtained using standardized equipment and protocols established previously in the CRIC Study. Blood and urine samples will be collected for serum creatinine, serum cystatin C, and urine protein/creatinine, the key indicators of kidney outcomes. Serum creatinine will be measured locally using CLIA-approved laboratories, and serum cystatin C and urine protein/creatinine will be measured at the CRIC Central Laboratory (CCL) at the University of Pennsylvania. As has been done in earlier phases, the results of the serum creatinine measurement will be provided to participants. Serum and urine remaining after the centralized measurements will be stored at the CCL during the Phase 5 award period for potential analyses in the future. For participants who are unable to come to the Clinical Center for an in-person visit, informed consent and the medical history and hospitalization data will be obtained by telephone. Participants should be encouraged to get blood drawn at a laboratory or at their home if they are not able to come to the Clinical Center.

Phase 5 Visit 2

The follow-up visit for participants without ESKD can take place by telephone or in person. During the follow-up visit, medical history updates and hospitalization data will be collected.

The subset of participants who participated in any of the three Phase 4 subprotocols will be asked to have a second blood draw for creatinine measurement at or around the time of Visit 2. The creatinine measurement can be performed at the study site, at a commercial laboratory, or at the participant's home.

Follow-up of Participants who have Reached ESKD

Participants who have reached ESKD before the start of Phase 5 will not have in person visits but will be consented via a telephone visit for passive follow-up through linkages with the US Renal Data System, the National Death Index, and other national billing claims or other databases. These participants will also be asked to consent to sharing their contact information with the SDCC to facilitate potential future studies. Sharing of contact information is not required for participation in Phase 5. While participants who have reached ESKD will not undergo in-person visits as part of the core CRIC Phase 5 protocol, they may be invited to complete additional visits/activities for ancillary studies.

Close Out Activities

During the 3 years of the Clinical Center Phase 5 funding period, the Clinical Centers will hold local events to express appreciation to study participants for their contribution over many years and to provide them with an overview of major findings. The last 6 months of the Clinical Center funding period will focus on closeout activities including resolution of data queries, storage of study documents, and regulatory reporting and completion of outcome ascertainment.

ELIGIBILITY:
Inclusion Criteria:

During the screening visit a blood sample will be tested to indirectly check kidney function based on the serum creatinine level:

* Age Range: 21 - 79 years
* Estimated Glomerular Filtration Rate (GFR): 45 - 70 mL/min/1.73m²
* Proteinuria: varies dependent on eGRF

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Previously received dialysis (peritoneal and/or hemodialysis) lasting more than one month
* Prior organ or bone marrow transplant
* Prior renal transplant
* Received immunosuppressive or other immunotherapy for primary renal disease or systemic vasculitis that affects the kidneys (i.e., anti-GCM, ANCA, SLE, IgA nephropathy, cryoglobulin, etc.) within the past six months before enrollment
* Received chemotherapy or alkylating agents for systemic cancer
* Known cirrhosis
* NYHA Class III or IV heart failure at baseline
* Previous diagnosis of multiple myeloma or renal carcinoma
* Previously diagnosed polycystic kidney disease
* Known HIV infection and/or AIDS
* Pregnant or breast-feeding women
* Currently participating in an interventional clinical trial (i.e., primarily trials of therapeutic agents that may have an effect on renal or cardiovascular outcomes).
* Institutionalized (e.g., prisoner, nursing home resident, skilled nursing facility resident)
* Appears unlikely or unable to participate in the required study procedures as assessed by the investigator, study coordinator or designee.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Phase I of the CRIC Study a total of 3,939 individuals across the spectrum of severity of kidney disease were enrolled to ensure that a sufficient number of patients reach the primary study endpoints of kidney disease progression and cardiovascular events. During CRIC Phase III, an additional 1,560 older participants with milder severity of kidney disease were recruited. The 1,560 new cohort members, compared with participants recruited in Phase I, have higher ranges of age and more preserved kidney function, and most have proteinuria. The population of 1560 new recruits have similar characteristics as the current CRIC cohort: ~50% with Diabetes, ~50% female, ~45% white and ~45% African-American.
Sampling Method: Probability Sample
Enrollment: 5499 (Estimated)
Dates: Start 2003-07; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The slope of GFR is the primary outcome; Primary outcomes regarding CVD will focus on clinical events indicative of ischemic heart disease, CHF, stroke, and peripheral vascular disease supplemented by radiographic evidence of progressive CVD | 5 yrs

SECONDARY OUTCOMES:
1.Onset of ESRD; 2.Significant loss of renal function; 3.Composite clinical outcome defined by the occurrence of either 50% decline, or 25 l/min/1.73 m2 decline in GFR from baseline, or onset of ESRD; 4. Slope of change in proteinuria over time. | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dember, M.D., Study Director — University of Pennsylvania
Locations (12):
- United States (12):
  - Kaiser Permanente of Northern California, Oakland, California
  - University of California, San Francisco, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Wayne State - Harper University Hospital, Detroit, Michigan
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Feldman HI, Appel LJ, Chertow GM, Cifelli D, Cizman B, Daugirdas J, Fink JC, Franklin-Becker ED, Go AS, Hamm LL, He J, Hostetter T, Hsu CY, Jamerson K, Joffe M, Kusek JW, Landis JR, Lash JP, Miller ER, Mohler ER 3rd, Muntner P, Ojo AO, Rahman M, Townsend RR, Wright JT; Chronic Renal Insufficiency Cohort (CRIC) Study Investigators. The Chronic Renal Insufficiency Cohort (CRIC) Study: Design and Methods. J Am Soc Nephrol. 2003 Jul;14(7 Suppl 2):S148-53. doi: 10.1097/01.asn.0000070149.78399.ce. PMID 12819321
- [Background] Wimmer NJ, Townsend RR, Joffe MM, Lash JP, Go AS; Chronic Renal Insufficiency Cohort Study Investigators. Correlation between pulse wave velocity and other measures of arterial stiffness in chronic kidney disease. Clin Nephrol. 2007 Sep;68(3):133-43. PMID 17915615
- [Background] Stevens LA, Coresh J, Feldman HI, Greene T, Lash JP, Nelson RG, Rahman M, Deysher AE, Zhang YL, Schmid CH, Levey AS. Evaluation of the modification of diet in renal disease study equation in a large diverse population. J Am Soc Nephrol. 2007 Oct;18(10):2749-57. doi: 10.1681/ASN.2007020199. Epub 2007 Sep 12. PMID 17855641
- [Result] Xie D, Joffe MM, Brunelli SM, Beck G, Chertow GM, Fink JC, Greene T, Hsu CY, Kusek JW, Landis R, Lash J, Levey AS, O'Conner A, Ojo A, Rahman M, Townsend RR, Wang H, Feldman HI. A comparison of change in measured and estimated glomerular filtration rate in patients with nondiabetic kidney disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1332-8. doi: 10.2215/CJN.05631207. Epub 2008 Jul 30. PMID 18667734
- [Result] Lash JP, Go AS, Appel LJ, He J, Ojo A, Rahman M, Townsend RR, Xie D, Cifelli D, Cohan J, Fink JC, Fischer MJ, Gadegbeku C, Hamm LL, Kusek JW, Landis JR, Narva A, Robinson N, Teal V, Feldman HI; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Chronic Renal Insufficiency Cohort (CRIC) Study: baseline characteristics and associations with kidney function. Clin J Am Soc Nephrol. 2009 Aug;4(8):1302-11. doi: 10.2215/CJN.00070109. Epub 2009 Jun 18. PMID 19541818
- [Result] DeLoach SS, Appel LJ, Chen J, Joffe MM, Gadegbeku CA, Mohler ER 3rd, Parsa A, Perumal K, Rafey MA, Steigerwalt SP, Teal V, Townsend RR, Rosas SE. Aortic pulse pressure is associated with carotid IMT in chronic kidney disease: report from Chronic Renal Insufficiency Cohort. Am J Hypertens. 2009 Dec;22(12):1235-41. doi: 10.1038/ajh.2009.156. Epub 2009 Sep 24. PMID 19779470
- [Result] Muntner P, Anderson A, Charleston J, Chen Z, Ford V, Makos G, O'Connor A, Perumal K, Rahman M, Steigerwalt S, Teal V, Townsend R, Weir M, Wright JT Jr; Chronic Renal Insufficiency Cohort (CRIC) Study Investigators. Hypertension awareness, treatment, and control in adults with CKD: results from the Chronic Renal Insufficiency Cohort (CRIC) Study. Am J Kidney Dis. 2010 Mar;55(3):441-51. doi: 10.1053/j.ajkd.2009.09.014. Epub 2009 Dec 5. PMID 19962808
- [Result] Joffe M, Hsu CY, Feldman HI, Weir M, Landis JR, Hamm LL; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Variability of creatinine measurements in clinical laboratories: results from the CRIC study. Am J Nephrol. 2010;31(5):426-34. doi: 10.1159/000296250. Epub 2010 Apr 14. PMID 20389058
- [Result] Yaffe K, Ackerson L, Kurella Tamura M, Le Blanc P, Kusek JW, Sehgal AR, Cohen D, Anderson C, Appel L, Desalvo K, Ojo A, Seliger S, Robinson N, Makos G, Go AS; Chronic Renal Insufficiency Cohort Investigators. Chronic kidney disease and cognitive function in older adults: findings from the chronic renal insufficiency cohort cognitive study. J Am Geriatr Soc. 2010 Feb;58(2):338-45. doi: 10.1111/j.1532-5415.2009.02670.x. Epub 2010 Jan 26. PMID 20374407
- [Result] Townsend RR, Wimmer NJ, Chirinos JA, Parsa A, Weir M, Perumal K, Lash JP, Chen J, Steigerwalt SP, Flack J, Go AS, Rafey M, Rahman M, Sheridan A, Gadegbeku CA, Robinson NA, Joffe M. Aortic PWV in chronic kidney disease: a CRIC ancillary study. Am J Hypertens. 2010 Mar;23(3):282-9. doi: 10.1038/ajh.2009.240. Epub 2009 Dec 17. PMID 20019670
- [Result] Gutierrez OM, Anderson C, Isakova T, Scialla J, Negrea L, Anderson AH, Bellovich K, Chen J, Robinson N, Ojo A, Lash J, Feldman HI, Wolf M; CRIC Study Group. Low socioeconomic status associates with higher serum phosphate irrespective of race. J Am Soc Nephrol. 2010 Nov;21(11):1953-60. doi: 10.1681/ASN.2010020221. Epub 2010 Sep 16. PMID 20847142
- [Result] Grunwald JE, Alexander J, Maguire M, Whittock R, Parker C, McWilliams K, Lo JC, Townsend R, Gadegbeku CA, Lash JP, Fink JC, Rahman M, Feldman H, Kusek J, Ojo A; CRIC Study Group. Prevalence of ocular fundus pathology in patients with chronic kidney disease. Clin J Am Soc Nephrol. 2010 May;5(5):867-73. doi: 10.2215/CJN.08271109. Epub 2010 Mar 18. PMID 20299372
- [Result] Soliman EZ, Prineas RJ, Go AS, Xie D, Lash JP, Rahman M, Ojo A, Teal VL, Jensvold NG, Robinson NL, Dries DL, Bazzano L, Mohler ER, Wright JT, Feldman HI; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Chronic kidney disease and prevalent atrial fibrillation: the Chronic Renal Insufficiency Cohort (CRIC). Am Heart J. 2010 Jun;159(6):1102-7. doi: 10.1016/j.ahj.2010.03.027. PMID 20569726
- [Result] Townsend RR, Chirinos JA, Parsa A, Weir MA, Sozio SM, Lash JP, Chen J, Steigerwalt SP, Go AS, Hsu CY, Rafey M, Wright JT Jr, Duckworth MJ, Gadegbeku CA, Joffe MP; Chronic Renal Insufficiency Cohort Investigators. Central pulse pressure in chronic kidney disease: a chronic renal insufficiency cohort ancillary study. Hypertension. 2010 Sep;56(3):518-24. doi: 10.1161/HYPERTENSIONAHA.110.153924. Epub 2010 Jul 26. PMID 20660819
- [Result] Townsend RR, Anderson AH, Chen J, Gadebegku CA, Feldman HI, Fink JC, Go AS, Joffe M, Nessel LA, Ojo A, Rader DJ, Reilly MP, Teal V, Teff K, Wright JT, Xie D. Metabolic syndrome, components, and cardiovascular disease prevalence in chronic kidney disease: findings from the Chronic Renal Insufficiency Cohort (CRIC) Study. Am J Nephrol. 2011;33(6):477-84. doi: 10.1159/000327618. Epub 2011 Apr 27. PMID 21525746
- [Result] Kurella Tamura M, Xie D, Yaffe K, Cohen DL, Teal V, Kasner SE, Messe SR, Sehgal AR, Kusek J, DeSalvo KB, Cornish-Zirker D, Cohan J, Seliger SL, Chertow GM, Go AS. Vascular risk factors and cognitive impairment in chronic kidney disease: the Chronic Renal Insufficiency Cohort (CRIC) study. Clin J Am Soc Nephrol. 2011 Feb;6(2):248-56. doi: 10.2215/CJN.02660310. Epub 2010 Oct 7. PMID 20930087
- [Result] Hsu CY, Propert K, Xie D, Hamm L, He J, Miller E, Ojo A, Shlipak M, Teal V, Townsend R, Weir M, Wilson J, Feldman H; CRIC Investigators. Measured GFR does not outperform estimated GFR in predicting CKD-related complications. J Am Soc Nephrol. 2011 Oct;22(10):1931-7. doi: 10.1681/ASN.2010101077. Epub 2011 Sep 15. PMID 21921144
- [Result] Shlipak MG, Lash JP, Yang W, Teal V, Keane M, Cappola T, Keller C, Jamerson K, Kusek J, Delafontaine P, He J, Miller ER 3rd, Schreiber M, Go AS; CRIC Investigators. Symptoms characteristic of heart failure among CKD patients without diagnosed heart failure. J Card Fail. 2011 Jan;17(1):17-23. doi: 10.1016/j.cardfail.2010.08.009. PMID 21187260
- [Result] Isakova T, Anderson CA, Leonard MB, Xie D, Gutierrez OM, Rosen LK, Theurer J, Bellovich K, Steigerwalt SP, Tang I, Anderson AH, Townsend RR, He J, Feldman HI, Wolf M; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Diuretics, calciuria and secondary hyperparathyroidism in the Chronic Renal Insufficiency Cohort. Nephrol Dial Transplant. 2011 Apr;26(4):1258-65. doi: 10.1093/ndt/gfr026. Epub 2011 Mar 7. PMID 21382989
- [Result] Weir MR, Townsend RR, Fink JC, Teal V, Anderson C, Appel L, Chen J, He J, Litbarg N, Ojo A, Rahman M, Rosen L, Sozio SM, Steigerwalt S, Strauss L, Joffe MM. Hemodynamic correlates of proteinuria in chronic kidney disease. Clin J Am Soc Nephrol. 2011 Oct;6(10):2403-10. doi: 10.2215/CJN.01670211. Epub 2011 Aug 18. PMID 21852669
- [Result] Fischer MJ, Go AS, Lora CM, Ackerson L, Cohan J, Kusek JW, Mercado A, Ojo A, Ricardo AC, Rosen LK, Tao K, Xie D, Feldman HI, Lash JP; CRIC and H-CRIC Study Groups. CKD in Hispanics: Baseline characteristics from the CRIC (Chronic Renal Insufficiency Cohort) and Hispanic-CRIC Studies. Am J Kidney Dis. 2011 Aug;58(2):214-27. doi: 10.1053/j.ajkd.2011.05.010. Epub 2011 Jun 25. PMID 21705121
- [Result] Budoff MJ, Rader DJ, Reilly MP, Mohler ER 3rd, Lash J, Yang W, Rosen L, Glenn M, Teal V, Feldman HI; CRIC Study Investigators. Relationship of estimated GFR and coronary artery calcification in the CRIC (Chronic Renal Insufficiency Cohort) Study. Am J Kidney Dis. 2011 Oct;58(4):519-26. doi: 10.1053/j.ajkd.2011.04.024. Epub 2011 Jul 23. PMID 21783289
- [Result] Scialla JJ, Leonard MB, Townsend RR, Appel L, Wolf M, Budoff MJ, Chen J, Lustigova E, Gadegbeku CA, Glenn M, Hanish A, Raj D, Rosas SE, Seliger SL, Weir MR, Parekh RS; CRIC Study Group. Correlates of osteoprotegerin and association with aortic pulse wave velocity in patients with chronic kidney disease. Clin J Am Soc Nephrol. 2011 Nov;6(11):2612-9. doi: 10.2215/CJN.03910411. Epub 2011 Sep 22. PMID 21940840
- [Result] Ricardo AC, Lash JP, Fischer MJ, Lora CM, Budoff M, Keane MG, Kusek JW, Martinez M, Nessel L, Stamos T, Ojo A, Rahman M, Soliman EZ, Yang W, Feldman HI, Go AS; CRIC and HCRIC Investigators. Cardiovascular disease among hispanics and non-hispanics in the chronic renal insufficiency cohort (CRIC) study. Clin J Am Soc Nephrol. 2011 Sep;6(9):2121-31. doi: 10.2215/CJN.11341210. PMID 21896829
- [Result] Isakova T, Wahl P, Vargas GS, Gutierrez OM, Scialla J, Xie H, Appleby D, Nessel L, Bellovich K, Chen J, Hamm L, Gadegbeku C, Horwitz E, Townsend RR, Anderson CA, Lash JP, Hsu CY, Leonard MB, Wolf M. Fibroblast growth factor 23 is elevated before parathyroid hormone and phosphate in chronic kidney disease. Kidney Int. 2011 Jun;79(12):1370-8. doi: 10.1038/ki.2011.47. Epub 2011 Mar 9. PMID 21389978
- [Result] Faul C, Amaral AP, Oskouei B, Hu MC, Sloan A, Isakova T, Gutierrez OM, Aguillon-Prada R, Lincoln J, Hare JM, Mundel P, Morales A, Scialla J, Fischer M, Soliman EZ, Chen J, Go AS, Rosas SE, Nessel L, Townsend RR, Feldman HI, St John Sutton M, Ojo A, Gadegbeku C, Di Marco GS, Reuter S, Kentrup D, Tiemann K, Brand M, Hill JA, Moe OW, Kuro-O M, Kusek JW, Keane MG, Wolf M. FGF23 induces left ventricular hypertrophy. J Clin Invest. 2011 Nov;121(11):4393-408. doi: 10.1172/JCI46122. Epub 2011 Oct 10. PMID 21985788
- [Result] Isakova T, Xie H, Yang W, Xie D, Anderson AH, Scialla J, Wahl P, Gutierrez OM, Steigerwalt S, He J, Schwartz S, Lo J, Ojo A, Sondheimer J, Hsu CY, Lash J, Leonard M, Kusek JW, Feldman HI, Wolf M; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Fibroblast growth factor 23 and risks of mortality and end-stage renal disease in patients with chronic kidney disease. JAMA. 2011 Jun 15;305(23):2432-9. doi: 10.1001/jama.2011.826. PMID 21673295
- [Result] Anderson AH, Yang W, Hsu CY, Joffe MM, Leonard MB, Xie D, Chen J, Greene T, Jaar BG, Kao P, Kusek JW, Landis JR, Lash JP, Townsend RR, Weir MR, Feldman HI; CRIC Study Investigators. Estimating GFR among participants in the Chronic Renal Insufficiency Cohort (CRIC) Study. Am J Kidney Dis. 2012 Aug;60(2):250-61. doi: 10.1053/j.ajkd.2012.04.012. Epub 2012 Jun 2. PMID 22658574
- [Result] He J, Reilly M, Yang W, Chen J, Go AS, Lash JP, Rahman M, DeFilippi C, Gadegbeku C, Kanthety R, Tao K, Hamm LL, Ojo A, Townsend R, Budoff M; CRIC Investigators. Risk factors for coronary artery calcium among patients with chronic kidney disease (from the Chronic Renal Insufficiency Cohort Study). Am J Cardiol. 2012 Dec 15;110(12):1735-41. doi: 10.1016/j.amjcard.2012.07.044. Epub 2012 Sep 14. PMID 22980963
- [Result] Fischer MJ, Xie D, Jordan N, Kop WJ, Krousel-Wood M, Kurella Tamura M, Kusek JW, Ford V, Rosen LK, Strauss L, Teal VL, Yaffe K, Powe NR, Lash JP; CRIC Study Group Investigators. Factors associated with depressive symptoms and use of antidepressant medications among participants in the Chronic Renal Insufficiency Cohort (CRIC) and Hispanic-CRIC Studies. Am J Kidney Dis. 2012 Jul;60(1):27-38. doi: 10.1053/j.ajkd.2011.12.033. Epub 2012 Apr 11. PMID 22497791
- [Result] Chen J, Mohler ER 3rd, Xie D, Shlipak MG, Townsend RR, Appel LJ, Raj DS, Ojo AO, Schreiber MJ, Strauss LF, Zhang X, Wang X, He J, Hamm LL; CRIC Investigators. Risk factors for peripheral arterial disease among patients with chronic kidney disease. Am J Cardiol. 2012 Jul 1;110(1):136-41. doi: 10.1016/j.amjcard.2012.02.061. Epub 2012 Mar 31. PMID 22465315
- [Result] Adeseun GA, Xie D, Wang X, Joffe MM, Mohler ER 3rd, Townsend RR, Budoff M, Rosas SE. Carotid plaque, carotid intima-media thickness, and coronary calcification equally discriminate prevalent cardiovascular disease in kidney disease. Am J Nephrol. 2012;36(4):342-7. doi: 10.1159/000342794. Epub 2012 Sep 26. PMID 23107930
- [Result] Wahl P, Xie H, Scialla J, Anderson CA, Bellovich K, Brecklin C, Chen J, Feldman H, Gutierrez OM, Lash J, Leonard MB, Negrea L, Rosas SE, Anderson AH, Townsend RR, Wolf M, Isakova T; Chronic Renal Insufficiency Cohort Study Group. Earlier onset and greater severity of disordered mineral metabolism in diabetic patients with chronic kidney disease. Diabetes Care. 2012 May;35(5):994-1001. doi: 10.2337/dc11-2235. Epub 2012 Mar 23. PMID 22446176
- [Result] Lora CM, Ricardo AC, Brecklin CS, Fischer MJ, Rosman RT, Carmona E, Lopez A, Balaram M, Nessel L, Tao KK, Xie D, Kusek JW, Go AS, Lash JP. Recruitment of Hispanics into an observational study of chronic kidney disease: the Hispanic Chronic Renal Insufficiency Cohort Study experience. Contemp Clin Trials. 2012 Nov;33(6):1238-44. doi: 10.1016/j.cct.2012.07.012. Epub 2012 Jul 27. PMID 22841929
- [Result] Grunwald JE, Alexander J, Ying GS, Maguire M, Daniel E, Whittock-Martin R, Parker C, McWilliams K, Lo JC, Go A, Townsend R, Gadegbeku CA, Lash JP, Fink JC, Rahman M, Feldman H, Kusek JW, Xie D, Jaar BG; CRIC Study Group. Retinopathy and chronic kidney disease in the Chronic Renal Insufficiency Cohort (CRIC) study. Arch Ophthalmol. 2012 Sep;130(9):1136-44. doi: 10.1001/archophthalmol.2012.1800. PMID 22965589
- [Result] Grunwald JE, Ying GS, Maguire M, Pistilli M, Daniel E, Alexander J, Whittock-Martin R, Parker C, Mohler E, Lo JC, Townsend R, Gadegbeku CA, Lash JP, Fink JC, Rahman M, Feldman H, Kusek JW, Xie D, Coleman M, Keane MG; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Association between retinopathy and cardiovascular disease in patients with chronic kidney disease (from the Chronic Renal Insufficiency Cohort [CRIC] Study). Am J Cardiol. 2012 Jul 15;110(2):246-53. doi: 10.1016/j.amjcard.2012.03.014. Epub 2012 Apr 18. PMID 22516527
- [Result] Scialla JJ, Appel LJ, Wolf M, Yang W, Zhang X, Sozio SM, Miller ER 3rd, Bazzano LA, Cuevas M, Glenn MJ, Lustigova E, Kallem RR, Porter AC, Townsend RR, Weir MR, Anderson CA; Chronic Renal Insufficiency Cohort-CRIC Study Group. Plant protein intake is associated with fibroblast growth factor 23 and serum bicarbonate levels in patients with chronic kidney disease: the Chronic Renal Insufficiency Cohort study. J Ren Nutr. 2012 Jul;22(4):379-388.e1. doi: 10.1053/j.jrn.2012.01.026. Epub 2012 Apr 4. PMID 22480598
- [Result] Weir MR, Townsend RR, Fink JC, Teal V, Sozio SM, Anderson CA, Appel LJ, Turban S, Chen J, He J, Litbarg N, Ojo A, Rahman M, Rosen L, Steigerwalt S, Strauss L, Joffe MM. Urinary sodium is a potent correlate of proteinuria: lessons from the chronic renal insufficiency cohort study. Am J Nephrol. 2012;36(5):397-404. doi: 10.1159/000342966. Epub 2012 Oct 12. PMID 23076013
- [Result] Gupta J, Mitra N, Kanetsky PA, Devaney J, Wing MR, Reilly M, Shah VO, Balakrishnan VS, Guzman NJ, Girndt M, Periera BG, Feldman HI, Kusek JW, Joffe MM, Raj DS; CRIC Study Investigators. Association between albuminuria, kidney function, and inflammatory biomarker profile in CKD in CRIC. Clin J Am Soc Nephrol. 2012 Dec;7(12):1938-46. doi: 10.2215/CJN.03500412. Epub 2012 Sep 27. PMID 23024164
- [Result] Park M, Hsu CY, Li Y, Mishra RK, Keane M, Rosas SE, Dries D, Xie D, Chen J, He J, Anderson A, Go AS, Shlipak MG; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Associations between kidney function and subclinical cardiac abnormalities in CKD. J Am Soc Nephrol. 2012 Oct;23(10):1725-34. doi: 10.1681/ASN.2012020145. Epub 2012 Aug 30. PMID 22935481
- [Result] Yaffe K, Ackerson L, Hoang TD, Go AS, Maguire MG, Ying GS, Daniel E, Bazzano LA, Coleman M, Cohen DL, Kusek JW, Ojo A, Seliger S, Xie D, Grunwald JE; CRIC Study Investigators. Retinopathy and cognitive impairment in adults with CKD. Am J Kidney Dis. 2013 Feb;61(2):219-27. doi: 10.1053/j.ajkd.2012.10.006. Epub 2012 Dec 1. PMID 23206534
- [Result] Munoz Mendoza J, Isakova T, Ricardo AC, Xie H, Navaneethan SD, Anderson AH, Bazzano LA, Xie D, Kretzler M, Nessel L, Hamm LL, Negrea L, Leonard MB, Raj D, Wolf M; Chronic Renal Insufficiency Cohort. Fibroblast growth factor 23 and Inflammation in CKD. Clin J Am Soc Nephrol. 2012 Jul;7(7):1155-62. doi: 10.2215/CJN.13281211. Epub 2012 May 3. PMID 22554719
- [Result] Margolis DJ, Gupta J, Thom SR, Townsend RR, Kanetsky PA, Hoffstad O, Papdopoulos M, Fischer M, Schelling JR, Mitra N. Diabetes, lower extremity amputation, loss of protective sensation, and neuronal nitric oxide synthase associated protein in the chronic renal insufficiency cohort study. Wound Repair Regen. 2013 Jan-Feb;21(1):17-24. doi: 10.1111/j.1524-475X.2012.00866.x. Epub 2012 Dec 10. PMID 23228162
- [Result] Ricardo AC, Hacker E, Lora CM, Ackerson L, DeSalvo KB, Go A, Kusek JW, Nessel L, Ojo A, Townsend RR, Xie D, Ferrans CE, Lash JP; CRIC Investigators. Validation of the Kidney Disease Quality of Life Short Form 36 (KDQOL-36) US Spanish and English versions in a cohort of Hispanics with chronic kidney disease. Ethn Dis. 2013 Spring;23(2):202-9. PMID 23530302
- [Result] Bansal N, Keane M, Delafontaine P, Dries D, Foster E, Gadegbeku CA, Go AS, Hamm LL, Kusek JW, Ojo AO, Rahman M, Tao K, Wright JT, Xie D, Hsu CY; CRIC Study Investigators. A longitudinal study of left ventricular function and structure from CKD to ESRD: the CRIC study. Clin J Am Soc Nephrol. 2013 Mar;8(3):355-62. doi: 10.2215/CJN.06020612. Epub 2013 Feb 14. PMID 23411431
- [Result] Ferguson JF, Matthews GJ, Townsend RR, Raj DS, Kanetsky PA, Budoff M, Fischer MJ, Rosas SE, Kanthety R, Rahman M, Master SR, Qasim A, Li M, Mehta NN, Shen H, Mitchell BD, O'Connell JR, Shuldiner AR, Ho WK, Young R, Rasheed A, Danesh J, He J, Kusek JW, Ojo AO, Flack J, Go AS, Gadegbeku CA, Wright JT Jr, Saleheen D, Feldman HI, Rader DJ, Foulkes AS, Reilly MP; CRIC Study Principal Investigators. Candidate gene association study of coronary artery calcification in chronic kidney disease: findings from the CRIC study (Chronic Renal Insufficiency Cohort). J Am Coll Cardiol. 2013 Aug 27;62(9):789-98. doi: 10.1016/j.jacc.2013.01.103. Epub 2013 May 30. PMID 23727086
- [Result] Mishra RK, Li Y, DeFilippi C, Fischer MJ, Yang W, Keane M, Chen J, He J, Kallem R, Horwitz EJ, Rafey M, Raj DS, Go AS, Shlipak MG; CRIC Study Investigators. Association of cardiac troponin T with left ventricular structure and function in CKD. Am J Kidney Dis. 2013 May;61(5):701-9. doi: 10.1053/j.ajkd.2012.11.034. Epub 2013 Jan 4. PMID 23291148
- [Result] Mishra RK, Li Y, Ricardo AC, Yang W, Keane M, Cuevas M, Christenson R, deFilippi C, Chen J, He J, Kallem RR, Raj DS, Schelling JR, Wright J, Go AS, Shlipak MG; Chronic Renal Insufficiency Cohort Investigators. Association of N-terminal pro-B-type natriuretic peptide with left ventricular structure and function in chronic kidney disease (from the Chronic Renal Insufficiency Cohort [CRIC]). Am J Cardiol. 2013 Feb 1;111(3):432-8. doi: 10.1016/j.amjcard.2012.10.019. Epub 2012 Nov 22. PMID 23178053
- [Result] Scialla JJ, Lau WL, Reilly MP, Isakova T, Yang HY, Crouthamel MH, Chavkin NW, Rahman M, Wahl P, Amaral AP, Hamano T, Master SR, Nessel L, Chai B, Xie D, Kallem RR, Chen J, Lash JP, Kusek JW, Budoff MJ, Giachelli CM, Wolf M; Chronic Renal Insufficiency Cohort Study Investigators. Fibroblast growth factor 23 is not associated with and does not induce arterial calcification. Kidney Int. 2013 Jun;83(6):1159-68. doi: 10.1038/ki.2013.3. Epub 2013 Feb 6. PMID 23389416
- [Result] Liu KD, Yang W, Anderson AH, Feldman HI, Demirjian S, Hamano T, He J, Lash J, Lustigova E, Rosas SE, Simonson MS, Tao K, Hsu CY; Chronic Renal Insufficiency Cohort (CRIC) study investigators. Urine neutrophil gelatinase-associated lipocalin levels do not improve risk prediction of progressive chronic kidney disease. Kidney Int. 2013 May;83(5):909-14. doi: 10.1038/ki.2012.458. Epub 2013 Jan 23. PMID 23344473
- [Result] Dobre M, Yang W, Chen J, Drawz P, Hamm LL, Horwitz E, Hostetter T, Jaar B, Lora CM, Nessel L, Ojo A, Scialla J, Steigerwalt S, Teal V, Wolf M, Rahman M; CRIC Investigators. Association of serum bicarbonate with risk of renal and cardiovascular outcomes in CKD: a report from the Chronic Renal Insufficiency Cohort (CRIC) study. Am J Kidney Dis. 2013 Oct;62(4):670-8. doi: 10.1053/j.ajkd.2013.01.017. Epub 2013 Mar 13. PMID 23489677
- [Result] Ky B, Shults J, Keane MG, Sutton MS, Wolf M, Feldman HI, Reese PP, Anderson CA, Townsend RR, Deo R, Lo J, Gadegbeku C, Carlow D, Sulik MJ, Leonard MB; CRIC Study Investigators. FGF23 modifies the relationship between vitamin D and cardiac remodeling. Circ Heart Fail. 2013 Jul;6(4):817-24. doi: 10.1161/CIRCHEARTFAILURE.112.000105. Epub 2013 Jun 7. PMID 23748358
- [Derived] Dhamdhere R, Modanwal G, Mutha P, Medina S, Arepalli S, Rahman M, Al-Kindi S, Madabhushi A; CRIC Study Investigators. Fundus Photograph-Derived Computational Features Predict Risk of Cardiovascular Events in the Chronic Renal Insufficiency Cohort Clinical Observational Study. Kidney360. 2026 Jan 1;7(1):81-93. doi: 10.34067/KID.0000000955. Epub 2025 Aug 18. No abstract available. PMID 40824712
- [Derived] Park CH, Kim HW, Park JT, Chang TI, Yoo TH, Oh KH, Anderson AH, Yang W, Cohen JB, Rahman M, Kang SW, Han SH; on the behalf of CRIC Study and KNOW-CKD Investigators. BP and Kidney Disease Progression in Advanced CKD: Findings from the Chronic Renal Insufficiency Cohort and KoreaN Cohort Study for Outcome in Patients with CKD Studies. Clin J Am Soc Nephrol. 2025 Jun 6;20(9):1179-1189. doi: 10.2215/CJN.0000000760. PMID 40478754
- [Derived] Yuan Y, Liu M, Zhang S, Lin Y, Huang Y, Zhou H, Xu X, Zhuang X, Liao X. Effect of blood pressure index on clinical outcomes in patients with heart failure and chronic kidney disease. ESC Heart Fail. 2023 Dec;10(6):3330-3339. doi: 10.1002/ehf2.14437. Epub 2023 Sep 4. PMID 37667525
- [Derived] Anderson AH, Xie D, Wang X, Baudier RL, Orlandi P, Appel LJ, Dember LM, He J, Kusek JW, Lash JP, Navaneethan SD, Ojo A, Rahman M, Roy J, Scialla JJ, Sondheimer JH, Steigerwalt SP, Wilson FP, Wolf M, Feldman HI; CRIC Study Investigators. Novel Risk Factors for Progression of Diabetic and Nondiabetic CKD: Findings From the Chronic Renal Insufficiency Cohort (CRIC) Study. Am J Kidney Dis. 2021 Jan;77(1):56-73.e1. doi: 10.1053/j.ajkd.2020.07.011. Epub 2020 Aug 28. PMID 32866540
- [Derived] Anderson AH, Yang W, Townsend RR, Pan Q, Chertow GM, Kusek JW, Charleston J, He J, Kallem R, Lash JP, Miller ER 3rd, Rahman M, Steigerwalt S, Weir M, Wright JT Jr, Feldman HI; Chronic Renal Insufficiency Cohort Study Investigators. Time-updated systolic blood pressure and the progression of chronic kidney disease: a cohort study. Ann Intern Med. 2015 Feb 17;162(4):258-65. doi: 10.7326/M14-0488. PMID 25686166
- See also: The CRIC Study website has a section of general information about the study and kidney disease for members of the general public who may be interested. It includes a brief description of the study and the 13 participating clinical centers. — http://www.cristudy.org